CLINICAL TRIAL: NCT00616941
Title: A Phase 1 Study of NY-ESO-1 Overlapping Peptides With or Without Immunoadjuvants Montanide and Poly-ICLC Vaccination of Epithelial Ovarian Cancer, Fallopian Tube, or Primary Peritoneal Cancer Patients in Second or Third Remission
Brief Title: Phase 1 Study of NY-ESO-1 Overlapping Peptides in Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ludwig Institute for Cancer Research (Other)
Collaborators: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LUD2006-001; MSKCC IRB# 07-152
Record Dates: First submitted 2008-02-04; First posted 2008-02-15 (Estimated); Results first posted 2018-07-27 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Epithelial Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer
Keywords: NY-ESO-1 OLP4; Ovarian Cancer; Cancer Vaccine
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Monatide (IMS 3015); poly ICLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Subjects received 4 synthetic peptides coded by the NY-ESO-1 gene (ie, NY-ESO-1 OLP4) once every 3 weeks for a total of 5 vaccinations.
  Interventions: Biological: NY-ESO-1 OLP4
- Cohort 2 (Experimental): Subjects received 4 synthetic peptides coded by the NY-ESO-1 gene (ie, NY-ESO-1 OLP4) in combination with Montanide ISA-51 vegetable grade (VG) once every 3 weeks for a total of 5 vaccinations.
  Interventions: Biological: NY-ESO-1 OLP4 + Montanide
- Cohort 3 (Experimental): Subjects received 4 synthetic peptides coded by the NY-ESO-1 gene (ie, NY-ESO-1 OLP4) in combination with Montanide ISA-51 VG and poly-ICLC once every 3 weeks for a total of 5 vaccinations.
  Interventions: Biological: NY-ESO-1 OLP4 + Montanide + Poly-ICLC

INTERVENTIONS:
Biological: NY-ESO-1 OLP4 — 1.0 mg of NY-ESO-1 OLP4 (0.25 mg of each overlapping peptide) was diluted in 0.5 mL of 5% dextrose in water (D5W) and administered subcutaneously as a single injection.
  Arms: Cohort 1
Biological: NY-ESO-1 OLP4 + Montanide — 1.0 mg of NY-ESO-1 OLP4 (0.25 mg of each overlapping peptide) was diluted in 0.5 mL of D5W, mixed with 0.5 mL of Montanide, and administered subcutaneously as a single injection.
  Arms: Cohort 2
Biological: NY-ESO-1 OLP4 + Montanide + Poly-ICLC — 1.0 mg of NY-ESO-1 OLP4 (0.25 mg of each overlapping peptide) and 1.4 mg of poly-ICLC were emulsified in 1.0 mL of Montanide and administered subcutaneously as two injections.
  Arms: Cohort 3

SUMMARY:
This was a Phase 1, open-label study of repeated vaccination with NY-ESO-1 overlapping peptides (OLP4) with or without the immunoadjuvants Montanide and polyinosinic-polycytidylic acid - poly-L-lysine carboxymethylcellulose (poly-ICLC) administered every 3 weeks for a total of 5 vaccinations in subjects with epithelial ovarian, fallopian tube, or primary peritoneal cancer in second or third clinical remission. Study objectives included determination of the safety and immunogenicity following vaccination.

DETAILED DESCRIPTION:
Subjects received NY-ESO-1 OLP4 by subcutaneous injection once every 3 weeks (Weeks 1, 4, 7, 10, and 13) for a total of 5 vaccinations.

Subjects were assigned sequentially to 1 of 3 dosing cohorts:

Cohort 1: received NY-ESO-1 OLP4 alone; Cohort 2: received NY-ESO-1 OLP4 in combination with Montanide; Cohort 3: received NY-ESO-1 OLP4 in combination with Montanide and Poly-ICLC.

Enrollment into each subsequent dosing cohort was dependent on a dose-limiting toxicity (DLT) rate of <33% in the preceding cohort. No dose escalation was planned.

Subjects were observed by study staff for up to 30 minutes following each vaccination. Immunologic assessments were performed prior to the first vaccination and 3 weeks after each vaccination. Toxicity assessments were performed with each vaccination and 3 weeks after the completion of therapy (ie, the final study visit was Week 16). Immunologic assessments included measurement of the anti-NY-ESO-1 antibody by enzyme-linked immunsorbent assay (ELISA), detection of CD-4 and CD-8 cellular responses by tetramer and enzyme-linked immunosorbent spot assay (ELISPOT), and delayed-type hypersensitivity (DTH).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically documented epithelial carcinoma arising in the ovary, fallopian tube, or peritoneum, stage II to IV at diagnosis, and post-initial cytoreductive surgery and chemotherapy with at least one platinum-based chemotherapy regimen.
2. In second or third stable complete clinical remission, defined as a) stable cancer antigen (CA)-125 < 35 U/ml (defined as CA-125 that had not doubled from the post chemotherapy nadir), b) unremarkable physical examination, and c) no definite evidence of disease by computed tomography (CT) of the abdomen and pelvis. Lymph nodes and/or soft tissue abnormalities ≤ 1.0 cm that are often present in the pelvis were not considered definite evidence of disease.
3. Expected survival of at least 4 months.
4. Karnofsky performance scale ≥ 70%.
5. Laboratory values within the following limits:

   * Hemoglobin ≥ 10.0 g/dL
   * Neutrophil count ≥ 1.5 x 10^9/L
   * Platelet count ≥ 80 x 10^9/L
   * Serum creatinine ≤ 2.0 mg/dL
   * Serum bilirubin ≤ 2.5 x institutional upper limit of normal (ULN)
   * aspartate aminotransferase/alanine aminotransferase ≤ 2.5 x institutional ULN
6. Age ≥ 18 years.
7. ≥ 4 weeks since completion of prior cytotoxic chemotherapy.
8. Able and willing to give valid written informed consent

Exclusion Criteria:

1. Clinically significant heart disease (New York Heart Association Class III or IV).
2. Serious intercurrent illness, eg, serious infections requiring prolonged parenteral antibiotics or bleeding disorders requiring hospitalization.
3. Positive stool guaiac excluding hemorrhoids.
4. Known autoimmune disease (ie, rheumatoid arthritis, ulcerative colitis, etc); or immune deficiency (human immunodeficiency virus, hypogammaglobulinemia); or known active infections with Hepatitis B or Hepatitis C; or receipt of immunosuppressive drugs such as systemic corticosteroids or cyclosporin, etc.
5. Other malignancy within 3 years prior to entry into the study, except for treated non-melanoma skin cancer and cervical carcinoma in situ.
6. History of previous severe allergic reactions to vaccines or unknown allergens.
7. Mental impairment that may have compromised the ability to give informed consent and comply with the requirements of the study.
8. Lack of availability for immunological and clinical follow-up assessments.
9. Participation in any other clinical trial involving another investigational agent within 4 weeks prior to first dose of study agent.
10. Pregnancy or breast-feeding.
11. Women of childbearing potential: Refusal or inability to use effective means of contraception.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Subjects must have had selected female reproductive organ cancers.
Enrollment: 28 (Actual)
Dates: Start 2008-03 (Actual); Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Sabbatini, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data have been published

REFERENCES:
- [Result] Sabbatini P, Tsuji T, Ferran L, Ritter E, Sedrak C, Tuballes K, Jungbluth AA, Ritter G, Aghajanian C, Bell-McGuinn K, Hensley ML, Konner J, Tew W, Spriggs DR, Hoffman EW, Venhaus R, Pan L, Salazar AM, Diefenbach CM, Old LJ, Gnjatic S. Phase I trial of overlapping long peptides from a tumor self-antigen and poly-ICLC shows rapid induction of integrated immune response in ovarian cancer patients. Clin Cancer Res. 2012 Dec 1;18(23):6497-508. doi: 10.1158/1078-0432.CCR-12-2189. Epub 2012 Oct 2. PMID 23032745
- [Derived] Tsuji T, Sabbatini P, Jungbluth AA, Ritter E, Pan L, Ritter G, Ferran L, Spriggs D, Salazar AM, Gnjatic S. Effect of Montanide and poly-ICLC adjuvant on human self/tumor antigen-specific CD4+ T cells in phase I overlapping long peptide vaccine trial. Cancer Immunol Res. 2013 Nov;1(5):340-50. doi: 10.1158/2326-6066.CIR-13-0089. Epub 2013 Sep 16. PMID 24777970

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Subjects received 4 synthetic peptides coded by the NY-ESO-1 gene (ie, NY-ESO-1 overlapping peptides [OLP4]) once every 3 weeks for a total of 5 vaccinations.
  1.0 mg of NY-ESO-1 OLP4 (0.25 mg of each overlapping peptide) was diluted in 0.5 mL of 5% dextrose in water (D5W) and administered subcutaneously as a single injection.
- Cohort 2: Subjects received 4 synthetic peptides coded by the NY-ESO-1 gene (ie, NY-ESO-1 OLP4) in combination with Montanide ISA-51 vegetable grade (VG) once every 3 weeks for a total of 5 vaccinations.
  1.0 mg of NY-ESO-1 OLP4 (0.25 mg of each overlapping peptide) was diluted in 0.5 mL of D5W, mixed with 0.5 mL of Montanide, and administered subcutaneously as a single injection.
- Cohort 3: Subjects received 4 synthetic peptides coded by the NY-ESO-1 gene (ie, NY-ESO-1 OLP4) in combination with Montanide ISA-51 VG and polyinosinic-polycytidylic acid - poly-L-lysine carboxymethylcellulose (poly-ICLC) once every 3 weeks for a total of 5 vaccinations.
  1.0 mg of NY-ESO-1 OLP4 (0.25 mg of each overlapping peptide) and 1.4 mg of poly-ICLC were emulsified in 1.0 mL of Montanide and administered subcutaneously as two injections.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Started | 4 | 13 | 11
Completed | 3 | 8 | 5
Not Completed | 1 | 5 | 6
Not completed — Progressive Disease | 1 | 2 | 1
Not completed — Adverse Event | 0 | 1 | 1
Not completed — Subject Non-compliance | 0 | 0 | 1
Not completed — Unrelated Medical Illness/Complication | 0 | 2 | 0
Not completed — Vaccination Suspended | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Population: All Enrolled Subjects
Groups:
- Cohort 1: Subjects received 4 synthetic peptides coded by the NY-ESO-1 gene (ie, NY-ESO-1 OLP4) once every 3 weeks for a total of 5 vaccinations.
  1.0 mg of NY-ESO-1 OLP4 (0.25 mg of each overlapping peptide) was diluted in 0.5 mL of D5W and administered subcutaneously as a single injection.
- Cohort 2: Subjects received 4 synthetic peptides coded by the NY-ESO-1 gene (ie, NY-ESO-1 OLP4) in combination with Montanide ISA-51 VG once every 3 weeks for a total of 5 vaccinations.
  1.0 mg of NY-ESO-1 OLP4 (0.25 mg of each overlapping peptide) was diluted in 0.5 mL of D5W, mixed with 0.5 mL of Montanide, and administered subcutaneously as a single injection.
- Cohort 3: Subjects received 4 synthetic peptides coded by the NY-ESO-1 gene (ie, NY-ESO-1 OLP4) in combination with Montanide ISA-51 VG and poly-ICLC once every 3 weeks for a total of 5 vaccinations.
  1.0 mg of NY-ESO-1 OLP4 (0.25 mg of each overlapping peptide) and 1.4 mg of poly-ICLC were emulsified in 1.0 mL of Montanide and administered subcutaneously as two injections.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Total
Number analyzed (Participants) | 4 | 13 | 11 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (10.7) | 58.6 (7.7) | 57.1 (9.5) | 57.8 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 13 | 11 | 28
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 13 | 11 | 28
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 4 | 13 | 10 | 27
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 13 | 11 | 28
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 23.6 (4.8) | 29.1 (8.1) | 26.5 (6.6) | 27.3 (7.2)

OUTCOME MEASURES:

1. Primary Outcome: Overview of Treatment-emergent Adverse Events (TEAEs)
Description: Analysis of TEAEs reported from clinical laboratory tests, physical examinations, and vital signs from pre-treatment through 3 weeks after the last dose of study treatment.
Time Frame: Continuously for up to 16 weeks
Population: The Safety Analysis Set comprises all subjects who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 4 | 13 | 11
Participants
  Any TEAE | 3 | 13 | 11
  Treatment-related TEAE | 2 | 12 | 11
  TEAE Leading to Discontinuation | 0 | 3 | 1
  Dose-limiting toxicity | 0 | 1 | 0
  Serious TEAE | 0 | 1 | 0
  Death | 0 | 0 | 0

2. Secondary Outcome: Number of Patients With Detectable Serum Immunoglobulin G (IgG) Antibody Titers Against NY-ESO-1 Up to 16 Weeks Post-Baseline
Description: Blood samples were drawn to measure immunologic response at Screening and Weeks 4, 7, 10, 13, and 16. Specific antibodies against NY-ESO-1 were measured by enzyme-linked immunosorbent assay (ELISA).
Time Frame: Screening and Weeks 4, 7, 10, 13, and 16
Population: The Immune Response Analysis Set comprises all subjects who had available post-baseline results for a given immunologic measurement.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 4 | 13 | 11
Participants
  Detectable IgG Antibody Titers: Pretreatment | 1 | 0 | 1
  Detectable IgG Antibody Titers: Week 4 | 1 | 0 | 1
  Detectable IgG Antibody Titers: Week 7 | 1 | 0 | 7
  Detectable IgG Antibody Titers: Week 10 | 1 | 4 | 8
  Detectable IgG Antibody Titers: Week 13 | 1 | 4 | 8
  Detectable IgG Antibody Titers: Week 16 | 1 | 6 | 8

3. Secondary Outcome: Number of Patients With Detectable CD8+ and CD4+ T-cell Responses Up to 16 Weeks Post-Baseline
Description: Blood samples were drawn to measure immunologic response at Screening and Weeks 4, 7, 10, 13, and 16. NY-ESO-1-specific CD8+ and CD4+ T-cell reactivity was measured by tetramer analysis (in human leukocyte antigen [HLA] 0201* patients). Interferon gamma (IFN-γ) release by T cells was measured by the enzyme-linked immunospot (ELISPOT) assay. A subject was considered to have experienced a T-cell response if IFN-γ spots were detectable (>50 spots) by ELISPOT of 50,000 CD8+ and CD4+ T cells following pre-sensitization with a pool of 20-mer OLP covering all of NY-ESO-1 and tested against Epstein-Barr virus-transformed B cells pulsed with 3 subpools of these peptides.
Time Frame: Screening and Weeks 4, 7, 10, 13, and 16
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 4 | 13 | 11
Participants
  Any CD8 T-cell Response Post-Baseline | 1 | 9 | 10
  Any CD4 T-cell Response Post-Baseline | 4 | 13 | 11

4. Secondary Outcome: Number of Patients With Delayed-type Hypersensitivity (DTH) Reactions (Induration and Redness) to NY-ESO-1 OLP4 at Screening and Week 16
Description: NY-ESO-1-specific DTH was measured by skin tests at Screening and again at Week 16. NY-ESO-1 OLP4 (40 µg in 0.1 mL D5W) was injected intradermally, with DTH reactions read 48 hours after injection.
Time Frame: Screening and Week 16
Population: The Safety Analysis Set comprises all subjects who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 4 | 13 | 11
Participants
  Presence of Induration at Screening | 0 | 0 | 0
  Presence of Induration at Week 16 | 1 | 4 | 2
  Presence of Redness at Screening | 0 | 2 | 2
  Presence of Redness at Week 16 | 0 | 6 | 4

5. Secondary Outcome: Cancer Antigen (CA)-125 Levels Up to 16 Weeks Post-Baseline
Description: Serum CA-125 was measured at Screening, Week 7, and Week 16. Stable CA-125 at baseline was < 35 U/mL (defined as CA-125 that had not doubled from the post chemotherapy nadir).
Time Frame: Screening, Week 7, and Week 16
Population: The Tumor Response Analysis Set comprises all subjects who had a given post-baseline efficacy measurement performed.
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 4 | 13 | 11
U/mL
  Screening | 14.0 (12.7) | 8.5 (5.3) | 10.9 (4.4)
  Week 7 | 29.5 (44.3) | 13.8 (12.5) | 21.3 (25.8)
  Week 16 | 8.0 (1.0) | 12.9 (9.7) | 35.1 (66.0)

6. Secondary Outcome: Tumor Measurement Results According to the Response Evaluation Criteria for Solid Tumors (RECIST) Up to 16 Weeks Post-Baseline
Description: Radiographic imaging (computed tomography of the abdomen and pelvis) was obtained at Screening and every 2 months during the study, and at unscheduled time points if any clinical symptoms/examination findings warranted further evaluation or if serum CA-125 rose to > 70 U/mL (confirmed by repeat value). Subjects may have had more than 1 location of disease.
Time Frame: Screening and every 2 months up to Week 16
Population: The Tumor Response Analysis Set comprises all subjects who had a given post-baseline efficacy assessment performed.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 4 | 13 | 11
Participants
  Screening: Evidence of Disease | 0 | 0 | 0
  Week 7: Evidence of Disease | 1 | 0 | 1
  Week 7: Disease Location - Regional Lymph Node | 1 | 0 | 0
  Week 7: Disease Location - Liver | 0 | 0 | 1
  Week 7: Disease Location - Other | 0 | 0 | 1
  Week 16: Evidence of Disease | 0 | 4 | 1
  Week 16: Disease Location - Local Recurrence | 0 | 4 | 0
  Week 16: Disease Location - Liver | 0 | 1 | 1

ADVERSE EVENTS:
Time Frame: All AEs occurring between the signing of informed consent and the off-study date were documented, regardless of the causal relationship to study drug. AEs occurring after the first dose of study drug were considered treatment emergent (i.e., TEAEs). The AE reporting period for this study was up to 16 weeks for each subject.
Description: AE documentation included onset/resolution dates, severity using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) (version 3.0), frequency, seriousness, related interventions, and outcome. In summaries, treatment-related AEs included those with a "possible", "probable", or "definite" relationship to study drug; preferred terms were counted only once per subject at the maximum reported grade.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/13 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/13 | 0/11
Other Adverse Events (participants affected / at risk) | 3/4 | 13/13 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=4) | Cohort 2 (N=13) | Cohort 3 (N=11)
Pneumonia (Infections and infestations) | 0 | 1 | 0 — Grade 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=4) | Cohort 2 (N=13) | Cohort 3 (N=11)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1
Visual acuity reduced (Eye disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 4 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Injection site reaction (General disorders) | 1 | 7 | 10
Fatigue (General disorders) | 2 | 6 | 3
Injection site pain (General disorders) | 0 | 1 | 3
Pyrexia (General disorders) | 0 | 1 | 2
Influenza like illness (General disorders) | 0 | 2 | 0
Hernia (General disorders) | 0 | 1 | 0
Injection site erythema (General disorders) | 0 | 1 | 0
Injection site pruritus (General disorders) | 0 | 1 | 0
Injection site rash (General disorders) | 0 | 1 | 0
Oedema (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 3 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 3
Bronchitis (Infections and infestations) | 0 | 1 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood potassium decreased (Investigations) | 0 | 1 | 0
Neutrophil count abnormal (Investigations) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Panniculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin nodule (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less